CLINICAL TRIAL: NCT04010149
Title: The Impact of Concurrent Brain Stimulation and Working Memory Training on Cognitive Performance in Acquired Brain Injury
Brief Title: Computerised Working Memory Training in Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Northamptonshire Healthcare NHS Foundation Trust (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RG_18-142
Record Dates: First submitted 2019-06-27; First posted 2019-07-08 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-03

CONDITIONS: Acquired Brain Injury
Keywords: Working memory; cognitive training; tDCS
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Eligible participants will begin the administration of the baseline measures (T0), and outcome measures (T1). On the first training day, participants will receive active or sham brain stimulation, concurrent with one session of their training routine (20 minutes). Before each training session, participants will also be asked to answer short questions (level of alertness, engagement, etc.). Participants will complete 10 additional consecutive training sessions (2 weeks), at home. Each session should take about 45 minutes.
  When the first training phase is complete, the participant will undergo time 2 (T2) assessment, as in T1.
  Participants will then start the second training phase, involving 3 weeks of training only (no brain stimulation), at home. When the second training phase is completed, participants will undergo time 3 (T3) assessment, as in T2.
  A last follow-up assessment, as T3, will be carried out at T4, a month after the completion of the intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A computer programme will generate a random list assigning group allocation to participant numbers. The participant numbers will be given out in order of attendance in the laboratory. The study design is double blind: participants and the researchers who are conducting the behavioural testing will not know until the end of the intervention if the participant received brain stimulation. A researcher from the University of Birmingham (Dr Assecondi) will setup the blind protocol on the brain stimulation device and will keep a record of this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): During cognitive training in the first 2 weeks, participants will also received brain stimulation. The investigators will use a total current intensity of 2mA for 20 minutes, preceded by 30 seconds ramping up and followed by 30 seconds ramping down (total stimulation time = 21s).
  Interventions: Device: Active tDCS
- SHAM tDCS (Sham Comparator): During sham stimulation, concurrent with the cognitive training, The investigators will use the same setup as in the active condition but after ramping up, the current will be brought back to zero and the process repeated 30 seconds before the end of the 21 minutes time interval (total sham stimulation time = 21s).
  Interventions: Device: SHAM tDCS

INTERVENTIONS:
Device: Active tDCS — For the first two weeks of the study, participants will receive 20 min of brain stimulation, concurrent with cognitive training. Electrodes will be placed over the dorsolateral prefrontal cortex (active electrode), and the contralateral supraorbital site (return electrode).
  Arms: Active tDCS
Device: SHAM tDCS — For the first two weeks of the study, participants will receive 20 min of SHAM brain stimulation, concurrent with cognitive training. Electrodes will be placed over the dorsolateral prefrontal cortex (active electrode), and the contralateral supraorbital site (return electrode).
  Arms: SHAM tDCS

SUMMARY:
Working memory is a limited capacity cognitive system in which information is held temporarily in order to make it available for processing. The amount of information that can be held in mind varies considerably from person to person and changes across the lifespan.

Working memory is frequently affected following brain injury. As working memory is important for cognitive skills such as problem solving, planning and active listening, a deficit in working memory can lead to difficulties with many everyday activities that are necessary for work, study and general functioning. Impaired working memory may consequently have a significant impact on a person's quality of life and ability to participate in previous social roles, with potential for effects on mood and emotional wellbeing.

Evidence shows that non-invasive transcranial direct current brain stimulation (tDCS) can be used in combination with computerized memory training (CT) over multiple days, to enhance working memory in healthy and clinical populations. In patients with an acquired brain injury (ABI), cognitive training or brain stimulation have been used alone to improve attention or memory-related impairment, but the effect of the concurrent used of the two interventions over multiple days is yet to be investigated.

With this research the investigators propose to investigate the effect of the combined use of tDCS and CT to improve memory performance in patients with acquired brain injury. The investigators propose to use a multi-day cognitive training regime to exercise working memory, while stimulating the brain with low intensity direct currents. Success will be measured as improvement in performance in several cognitive domain, before and after training.

DETAILED DESCRIPTION:
Participants will be recruited through Northampton Healthcare NHS Foundation Trust Acquired Brain Injury clinics. They will complete 5 weeks of training at home. During the first two weeks they will be visited in their home by a researcher who will administered the current stimulation together with the working memory training program. The remaining 3 weeks the patient will complete the training program at home, while receiving a motivational / catch up call every week. Weekends will be exempt from testing. The working memory training software program is accessed via a password-protected website on a secure server at Dalhousie University. Training data will be saved on the Dalhousie University server and will be downloaded in Birmingham for data analyses.

RECRUITMENT As the aim of this research is to improve spatial working memory, only participants with a working memory impairment will be included in the study. To identify a working memory impairment, cognitive tests from the Wechsler Adult Intelligence Test (WAIS-IV) and the Wechsler Memory Scale (WMS-IV), will be administered in paper and pencil versions or using iPads. These tests are administered to every patient, as part of the routine care protocol.

The investigators will consider the following scores:

* A Full-Scale Intelligent Quotient (FSIQ) obtained from the WAIS-IV higher than 70: this score identifies patients able to follow instructions. The FSIQ will also be used as a covariate in the analysis to control for low average overall ability rather than a specific working memory issue.
* A Working Memory Index (WMI), obtained as a combination of the digit span score and the arithmetic score in the WAIS-IV, smaller than 85: this score identifies a general working memory impairment;
* A Visual Working Memory Index (VWMI), obtained as a combination of the symbol span and the spatial addition score in the WMS-IV, smaller than 85: this score identifies impairment specific to spatial working memory.

These tests are co-normed on a large sample (mean = 100; SD = 15). In order to be included in the study, a patient should have a FSIQ >70 and either a WMI or a SWMI or both < 85. This means that the investigators use a criterion score of one standard deviation below the mean. This score doesn't reflect significant impairment, but it allows us to identify patients with an impairment significant enough to potentially improve with training. See below for a detailed description of the cognitive tasks used. Participants who don't present a working memory impairment, as defined above, will be excluded from further participation. Patients identified as potential participants in the study will be approached with a letter.

SCREENING PROCEDURE:

Following the informed consent procedure, each participant will be randomly assigned to one of the two training conditions (active or sham stimulation) and interviewed with a Screening Questionnaire, which includes questions about demographic information and health history that will evaluate the inclusion/exclusion criteria. The investigators will also ask about current medications and information about time since injury, handedness and colour blindness will be recorded. At this point, participants who don't meet the eligibility criteria will be excluded from further participation. Finally, participants will be made aware of possible side effects of brain stimulation and they will ask to confirm their willingness to participate in the study.

TESTING AND TRAINING:

The protocol is detailed in the protocol flowchart (Annexe 5). After the consent and screening procedures, eligible participants will begin the administration of the baseline measures (T0), and outcome measures (T1). The baseline measures involve completing a series of questionnaires (see below for a list and a brief explanation of each questionnaire), since these variables may impact performance on the tasks. The baseline data will be included in our data analyses as potential modifiers of performance. In total, the investigators expect the entirety of the first in-lab session (informed consent, screening, and baseline measures (T0)) to take about 1 hour. In addition, participants will be asked to refrain from excessive alcohol or coffee drinking during the intervention and to maintain good sleeping habits, where possible. On the following day participants will perform a series of pre-training outcome tasks (see above) to measure their working memory capacity baseline (T1) and to assess, during and at the end of the training intervention, the efficacy of the training and the stimulation regime. Participants will then be offered a break before familiarizing them with the stimulation procedure (sham or active according to the group they belong to) and the training game. The trainer will answer any questions about the study. This second session will last for about 1 h. On T1, the cognitive screening measures (WAIS-IV and WMS-IV) will not be repeated, as already administered as part of the routine care.

On the first training day after the T1 session, depending on the group, participants will receive active or sham brain stimulation (see below for stimulation parameters). At the same time, both groups will complete one session of the NIGMA game, e.g., one session of their training routine (20 minutes). Before each training session, participants will also be asked to answer short questions (level of alertness, engagement, etc.). Once the training session and the stimulation are completed, the participant will fill in a feedback form on the experienced side effects of brain stimulation, if any.

Participants will complete 10 additional consecutive training sessions (2 weeks, excluding weekends). Each session should take about 45 minutes (~10 minutes setting up of tDCS and ~20 minutes of N-IGMA training). This phase will be completed at home, with the researcher visiting the participant at a convenient time.

When the first training phase is complete, the participant will undergo time 2 (T2) assessment. Like before, this involves completing a series of computerised cognitive tasks to measures training gains and transfer (see "outcome measures" section, including also WAIS-IV and WMS-IV).

Participants will then start the second training phase, involving 3 weeks of training only (no brain stimulation). During this phase, patients will stay at home and access the training program via internet. Manualised phone calls will be used to educate the patients about attention and how they could apply the training to their daily life, to promote generalisation. When the second training phase is completed, participants will undergo time 3 (T3) assessment, during which they will repeat the same series of computerised cognitive tasks as in T2.

A last follow-up assessment, identical to the one at T2, and T3, will be carried out at T4, a month after the completion of the intervention, to assess maintenance of working memory improvements and transfer.

BRAIN STIMULATION PROTOCOL The brain stimulation targets the right dorsolateral prefrontal cortex (DLPFC). A bipolar setup will be used. The bipolar setup includes two Ag/AgCl electrodes filled with conductive EEG gel and placed on F4 (active electrode) and Fp1(return electrode). Reference electrodes will be attached to the earlobe and impedances will be measured throughout the stimulation. If impedances exceed 20kOhm at any time, the stimulation will automatically stop and will not resume until impedances are restored. The investigators will use a total current intensity of 2mA for 20 minutes, preceded by 30 seconds ramping up and followed by 30 seconds ramping down (total stimulation time = 21s). With these parameters and Ag/AgCl electrodes (area 3.14 cm2) a current density of approximately 0.6 mA/cm^2 is obtained, slightly higher than the one obtained with larger electrodes, but still well below the threshold for tissue damage (Antal et al., 2017; Bikson et al., 2016; Liebetanz et al., 2009)). During sham stimulation the investigators will use the same setup as in the active condition but after ramping up, the current will be brought back to zero and the process repeated 30 seconds before the end of the 21 minutes time interval (total sham stimulation time = 21s).

DATA ANALYSIS The investigators will analyse the data using parametric statistics if appropriate. These will include mixed and repeated measures ANOVAs, with factors such as group and test variables. Significant main effects and interactions (p < .05) will be followed by post-hoc tests corrected for multiple comparisons. Dependent variables on the computerized tasks will include mean reaction time (RT) and accuracy (% correct).

ELIGIBILITY:
Inclusion Criteria:

1. Referred to the service
2. Are between 18 and 69 years of age
3. Have capacity and able to provide informed consent
4. Normal or corrected-to-normal vision and hearing
5. Having a working memory impairment (see screening procedure below)
6. At least three months between the injury and the starting of the study
7. Has a computer or has access to a computer

Exclusion Criteria:

1. Pre-injury psychiatric or neurological disease by self-report (e.g., anxiety disorder, ADHD, Parkinson's disease, etc.)
2. History of diagnosed severe depression (diagnosed pre-injury)
3. History of epilepsy (diagnosed pre-injury)
4. Family history of epilepsy
5. Have had fainting spells or syncope in the last three years pre-injury
6. Have significant hearing loss, vision or motor impairment that would prevent them from performing the task
7. Known to be pregnant
8. Assuming medication affecting cortical excitability or recreational drugs
9. Metal (except titanium) or electronic implants in the brain /skull (e.g., splinters, fragments, clips, cochlear implant, deep brain stimulation, medication pump…)
10. Metal (except titanium) or any electronic device at other sites in the participant's body, such as cardiac pacemaker or traumatic metallic residual fragments
11. Have skin problems such as dermatitis, psoriasis or eczema under the stimulation sites
12. Have had brain stimulation in the past six months
13. Have undergone transcranial electric or magnetic stimulation in the past (more than 6 months) which resulted in adverse effects
14. Skull fractures, significant skull defects, skull plates or large vessels occlusions in the site of electrode placement
15. having had a seizure at the time of accident or between the injury and starting of the therapy.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Changes in memory capacity, as measured by number of items that are memorised successfully, in the cognitive task used as the training regime; | On day1, at end of week 2, at end of week 5 and at end of week 9
  The difficulty of the training regime is manipulated by increasing N, i.e. the number of items the participant is requested to memorise. As such, N is used to measure individual memory capacity. Changes in memory capacity, as the training regime progresses is the primary outcome measure of this study.

SECONDARY OUTCOMES:
Changes in memory capacity, as measured by number of items that are memorised successfully, in untrained cognitive tasks. | On day1, at end of week 2, at end of week 5 and at end of week 9
  Changes in the number of items memorised successfully are measured in a task different from the training task, but that tap into the same cognitive process (near transfer), or from a different task tapping into a different cognitive domain (mid transfer).
Persistence of changes in memory capacity through time | On day1, at end of week 2, at end of week 5 and at end of week 9
  Maintenance of memory capacity changes after termination of the training, as measured by the memory capacity, i.e., number of items memorised successfully, at different time point during and a month after the completion of the intervention, with respect to day 1 of the intervention.

OTHER OUTCOMES:
Impact of the intervention on self-reported everyday cognitive perfomrance, as measured by the PRECiS questionnaire. | On day1, at end of week 2, at end of week 5 and at end of week 9
  Impact of the intervention on self-reported everyday cognitive performance as measured by the Patient Reported Evaluation of Cognitive Status (PRECiS), taken at different time points along and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kimron Shapiro, Principal Investigator — University of Birmingham

REFERENCES:
- [Background] Akerlund E, Esbjornsson E, Sunnerhagen KS, Bjorkdahl A. Can computerized working memory training improve impaired working memory, cognition and psychological health? Brain Inj. 2013;27(13-14):1649-57. doi: 10.3109/02699052.2013.830195. Epub 2013 Oct 2. PMID 24087909
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Au J, Katz B, Buschkuehl M, Bunarjo K, Senger T, Zabel C, Jaeggi SM, Jonides J. Enhancing Working Memory Training with Transcranial Direct Current Stimulation. J Cogn Neurosci. 2016 Sep;28(9):1419-32. doi: 10.1162/jocn_a_00979. Epub 2016 May 11. PMID 27167403
- [Background] Baddeley A. Working memory: theories, models, and controversies. Annu Rev Psychol. 2012;63:1-29. doi: 10.1146/annurev-psych-120710-100422. Epub 2011 Sep 27. PMID 21961947
- [Background] Barbey AK, Koenigs M, Grafman J. Dorsolateral prefrontal contributions to human working memory. Cortex. 2013 May;49(5):1195-205. doi: 10.1016/j.cortex.2012.05.022. Epub 2012 Jun 16. PMID 22789779
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Chiesa A, Calati R, Serretti A. Does mindfulness training improve cognitive abilities? A systematic review of neuropsychological findings. Clin Psychol Rev. 2011 Apr;31(3):449-64. doi: 10.1016/j.cpr.2010.11.003. Epub 2010 Dec 1. PMID 21183265
- [Background] Christodoulou C, DeLuca J, Ricker JH, Madigan NK, Bly BM, Lange G, Kalnin AJ, Liu WC, Steffener J, Diamond BJ, Ni AC. Functional magnetic resonance imaging of working memory impairment after traumatic brain injury. J Neurol Neurosurg Psychiatry. 2001 Aug;71(2):161-8. doi: 10.1136/jnnp.71.2.161. PMID 11459886
- [Background] Course-Choi J, Saville H, Derakshan N. The effects of adaptive working memory training and mindfulness meditation training on processing efficiency and worry in high worriers. Behav Res Ther. 2017 Feb;89:1-13. doi: 10.1016/j.brat.2016.11.002. Epub 2016 Nov 10. PMID 27838273
- [Background] Datta A, Bikson M, Fregni F. Transcranial direct current stimulation in patients with skull defects and skull plates: high-resolution computational FEM study of factors altering cortical current flow. Neuroimage. 2010 Oct 1;52(4):1268-78. doi: 10.1016/j.neuroimage.2010.04.252. Epub 2010 May 7. PMID 20435146
- [Background] Dunning DL, Westgate B, Adlam AR. A meta-analysis of working memory impairments in survivors of moderate-to-severe traumatic brain injury. Neuropsychology. 2016 Oct;30(7):811-819. doi: 10.1037/neu0000285. Epub 2016 May 16. PMID 27182710
- [Background] Elmasry J, Loo C, Martin D. A systematic review of transcranial electrical stimulation combined with cognitive training. Restor Neurol Neurosci. 2015;33(3):263-78. doi: 10.3233/RNN-140473. PMID 25624425
- [Background] Giordano J, Bikson M, Kappenman ES, Clark VP, Coslett HB, Hamblin MR, Hamilton R, Jankord R, Kozumbo WJ, McKinley RA, Nitsche MA, Reilly JP, Richardson J, Wurzman R, Calabrese E. Mechanisms and Effects of Transcranial Direct Current Stimulation. Dose Response. 2017 Feb 9;15(1):1559325816685467. doi: 10.1177/1559325816685467. eCollection 2017 Jan-Mar. PMID 28210202
- [Background] Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. Proc Natl Acad Sci U S A. 2008 May 13;105(19):6829-33. doi: 10.1073/pnas.0801268105. Epub 2008 Apr 28. PMID 18443283
- [Background] Jeon SY, Han SJ. Improvement of the working memory and naming by transcranial direct current stimulation. Ann Rehabil Med. 2012 Oct;36(5):585-95. doi: 10.5535/arm.2012.36.5.585. Epub 2012 Oct 31. PMID 23185722
- [Background] Jo JM, Kim YH, Ko MH, Ohn SH, Joen B, Lee KH. Enhancing the working memory of stroke patients using tDCS. Am J Phys Med Rehabil. 2009 May;88(5):404-9. doi: 10.1097/PHM.0b013e3181a0e4cb. PMID 19620953
- [Background] Jones SA, Butler BC, Kintzel F, Johnson A, Klein RM, Eskes GA. Measuring the Performance of Attention Networks with the Dalhousie Computerized Attention Battery (DalCAB): Methodology and Reliability in Healthy Adults. Front Psychol. 2016 Jun 7;7:823. doi: 10.3389/fpsyg.2016.00823. eCollection 2016. PMID 27375517
- [Background] Kang EK, Kim DY, Paik NJ. Transcranial direct current stimulation of the left prefrontal cortex improves attention in patients with traumatic brain injury: a pilot study. J Rehabil Med. 2012 Apr;44(4):346-50. doi: 10.2340/16501977-0947. PMID 22434324
- [Background] Klingberg T. Training and plasticity of working memory. Trends Cogn Sci. 2010 Jul;14(7):317-24. doi: 10.1016/j.tics.2010.05.002. Epub 2010 Jun 16. PMID 20630350
- [Background] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Background] Lindelov JK, Overgaard R, Overgaard M. Improving working memory performance in brain-injured patients using hypnotic suggestion. Brain. 2017 Apr 1;140(4):1100-1106. doi: 10.1093/brain/awx001. PMID 28335012
- [Background] Liu A, Bryant A, Jefferson A, Friedman D, Minhas P, Barnard S, Barr W, Thesen T, O'Connor M, Shafi M, Herman S, Devinsky O, Pascual-Leone A, Schachter S. Exploring the efficacy of a 5-day course of transcranial direct current stimulation (TDCS) on depression and memory function in patients with well-controlled temporal lobe epilepsy. Epilepsy Behav. 2016 Feb;55:11-20. doi: 10.1016/j.yebeh.2015.10.032. Epub 2015 Dec 22. PMID 26720704
- [Background] Lundqvist A, Grundstrom K, Samuelsson K, Ronnberg J. Computerized training of working memory in a group of patients suffering from acquired brain injury. Brain Inj. 2010;24(10):1173-83. doi: 10.3109/02699052.2010.498007. PMID 20715888
- [Background] Mameli, F., Fumagalli, M., Ferrucci, R., & Priori, A. (2014). The Stimulated Brain. PART III: IMPROVING FUNCTIONS IN THE ATYPICAL BRAIN, 371-395.
- [Background] Conway, A. R., Jarrold, C., Kane, M. J., Miyake, A., & Towse, J. N. (2008). Variation in Working Memory, 3-18.
- [Background] Manktelow AE, Menon DK, Sahakian BJ, Stamatakis EA. Working Memory after Traumatic Brain Injury: The Neural Basis of Improved Performance with Methylphenidate. Front Behav Neurosci. 2017 Apr 5;11:58. doi: 10.3389/fnbeh.2017.00058. eCollection 2017. PMID 28424597
- [Background] Nilsson J, Lebedev AV, Rydstrom A, Lovden M. Direct-Current Stimulation Does Little to Improve the Outcome of Working Memory Training in Older Adults. Psychol Sci. 2017 Jul;28(7):907-920. doi: 10.1177/0956797617698139. Epub 2017 May 16. PMID 28509625
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Nyberg L, Lovden M, Riklund K, Lindenberger U, Backman L. Memory aging and brain maintenance. Trends Cogn Sci. 2012 May;16(5):292-305. doi: 10.1016/j.tics.2012.04.005. PMID 22542563
- [Background] Passow S, Thurm F, Li SC. Activating Developmental Reserve Capacity Via Cognitive Training or Non-invasive Brain Stimulation: Potentials for Promoting Fronto-Parietal and Hippocampal-Striatal Network Functions in Old Age. Front Aging Neurosci. 2017 Feb 23;9:33. doi: 10.3389/fnagi.2017.00033. eCollection 2017. PMID 28280465
- [Background] Paulus W. Transcranial direct current stimulation (tDCS). Suppl Clin Neurophysiol. 2003;56:249-54. doi: 10.1016/s1567-424x(09)70229-6. PMID 14677402
- [Background] Perceval G, Floel A, Meinzer M. Can transcranial direct current stimulation counteract age-associated functional impairment? Neurosci Biobehav Rev. 2016 Jun;65:157-72. doi: 10.1016/j.neubiorev.2016.03.028. Epub 2016 Apr 2. PMID 27048962
- [Background] Rabinowitz AR, Levin HS. Cognitive sequelae of traumatic brain injury. Psychiatr Clin North Am. 2014 Mar;37(1):1-11. doi: 10.1016/j.psc.2013.11.004. Epub 2014 Jan 14. PMID 24529420
- [Background] Rolle CE, Anguera JA, Skinner SN, Voytek B, Gazzaley A. Enhancing Spatial Attention and Working Memory in Younger and Older Adults. J Cogn Neurosci. 2017 Sep;29(9):1483-1497. doi: 10.1162/jocn_a_01159. Epub 2017 Jun 27. PMID 28654361
- [Background] Ruf SP, Fallgatter AJ, Plewnia C. Augmentation of working memory training by transcranial direct current stimulation (tDCS). Sci Rep. 2017 Apr 21;7(1):876. doi: 10.1038/s41598-017-01055-1. PMID 28432349
- [Background] Sammer G, Reuter I, Hullmann K, Kaps M, Vaitl D. Training of executive functions in Parkinson's disease. J Neurol Sci. 2006 Oct 25;248(1-2):115-9. doi: 10.1016/j.jns.2006.05.028. Epub 2006 Jun 12. PMID 16765378
- [Background] Serino A, Ciaramelli E, Di Santantonio A, Malagu S, Servadei F, Ladavas E. Central executive system impairment in traumatic brain injury. Brain Inj. 2006 Jan;20(1):23-32. doi: 10.1080/02699050500309627. PMID 16403697
- [Background] Smith EE, Jonides J, Koeppe RA. Dissociating verbal and spatial working memory using PET. Cereb Cortex. 1996 Jan-Feb;6(1):11-20. doi: 10.1093/cercor/6.1.11. PMID 8670634
- [Background] Soveri A, Antfolk J, Karlsson L, Salo B, Laine M. Working memory training revisited: A multi-level meta-analysis of n-back training studies. Psychon Bull Rev. 2017 Aug;24(4):1077-1096. doi: 10.3758/s13423-016-1217-0. PMID 28116702
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Talsma LJ, Kroese HA, Slagter HA. Boosting Cognition: Effects of Multiple-Session Transcranial Direct Current Stimulation on Working Memory. J Cogn Neurosci. 2017 Apr;29(4):755-768. doi: 10.1162/jocn_a_01077. Epub 2016 Nov 29. PMID 27897670
- [Background] Thair H, Holloway AL, Newport R, Smith AD. Transcranial Direct Current Stimulation (tDCS): A Beginner's Guide for Design and Implementation. Front Neurosci. 2017 Nov 22;11:641. doi: 10.3389/fnins.2017.00641. eCollection 2017. PMID 29213226
- [Background] Toril P, Reales JM, Mayas J, Ballesteros S. Video Game Training Enhances Visuospatial Working Memory and Episodic Memory in Older Adults. Front Hum Neurosci. 2016 May 6;10:206. doi: 10.3389/fnhum.2016.00206. eCollection 2016. PMID 27199723
- [Background] van de Ven RM, Murre JM, Veltman DJ, Schmand BA. Computer-Based Cognitive Training for Executive Functions after Stroke: A Systematic Review. Front Hum Neurosci. 2016 Apr 20;10:150. doi: 10.3389/fnhum.2016.00150. eCollection 2016. PMID 27148007
- [Background] Villamar MF, Santos Portilla A, Fregni F, Zafonte R. Noninvasive brain stimulation to modulate neuroplasticity in traumatic brain injury. Neuromodulation. 2012 Jul;15(4):326-38. doi: 10.1111/j.1525-1403.2012.00474.x. Epub 2012 Jun 14. PMID 22882244
- [Background] Wager TD, Smith EE. Neuroimaging studies of working memory: a meta-analysis. Cogn Affect Behav Neurosci. 2003 Dec;3(4):255-74. doi: 10.3758/cabn.3.4.255. PMID 15040547
- [Background] Westerberg H, Jacobaeus H, Hirvikoski T, Clevberger P, Ostensson ML, Bartfai A, Klingberg T. Computerized working memory training after stroke--a pilot study. Brain Inj. 2007 Jan;21(1):21-9. doi: 10.1080/02699050601148726. PMID 17364516
- [Background] Yavari F, Jamil A, Mosayebi Samani M, Vidor LP, Nitsche MA. Basic and functional effects of transcranial Electrical Stimulation (tES)-An introduction. Neurosci Biobehav Rev. 2018 Feb;85:81-92. doi: 10.1016/j.neubiorev.2017.06.015. Epub 2017 Jul 6. PMID 28688701
- [Background] Zimerman M, Hummel FC. Non-invasive brain stimulation: enhancing motor and cognitive functions in healthy old subjects. Front Aging Neurosci. 2010 Dec 1;2:149. doi: 10.3389/fnagi.2010.00149. eCollection 2010. PMID 21151809
- [Derived] Assecondi S, Hu R, Eskes G, Read M, Griffiths C, Shapiro K. BRAINSTORMING: A study protocol for a randomised double-blind clinical trial to assess the impact of concurrent brain stimulation (tDCS) and working memory training on cognitive performance in Acquired Brain Injury (ABI). BMC Psychol. 2020 Nov 26;8(1):125. doi: 10.1186/s40359-020-00454-w. PMID 33243286